CLINICAL TRIAL: NCT05386550
Title: A Randomized, Double-blind, Placebo-controlled, 2-arm Phase III Study to Assess Efficacy and Safety of Xevinapant and Radiotherapy Compared to Placebo and Radiotherapy for Demonstrating Improvement of Disease-free Survival in Participants With Resected Squamous Cell Carcinoma of the Head and Neck, Who Are at High Risk for Relapse and Are Ineligible for High-dose Cisplatin (XRAY VISION)
Brief Title: Phase III Xevinapant (Debio 1143) and Radiotherapy in Resected LA SCCHN, High Risk, Cisplatin-ineligible Participants (XRAY VISION)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No major safety concerns were identified in the XRAY VISION study, however development program was discontinued due to the outcome of Phase III Trilynx study.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS202359_0002; 2022-001144-18 (EudraCT Number)
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer
Keywords: Adjuvant radiotherapy (RT); Stage III; Stage IVA; Stage IVB; Oral cavity; Oropharynx; Larynx; Hypopharynx; Unfit
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Diseases | interventions — N-benzhydryl-5-(2-(methylamino)propanamido)-3-(3-methylbutanoyl)-6-oxodecahydropyrrolo(1,2-a)(1,5)diazocine-8-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Xevinapant + IMRT (Experimental): Participants received 3 cycles of oral solution of Xevinapant at a dose of 200 milligrams per day (mg/day) once daily from Day 1 to 14, per 3-week cycle in combination with 66 Gray (Gy) of intensity modulated radiation therapy (IMRT) in 33 fractions, 2 Gy/fraction, 5 days/week followed by 3 cycles of monotherapy of Xevinapant at a dose of 200 mg/day from Day 1 to 14, per 3-week cycle (Each cycle is of 3 weeks).
  Interventions: Drug: Xevinapant; Radiation: IMRT
- Placebo + IMRT (Placebo Comparator): Participants received 3 cycles of oral solution of placebo matched to Xevinapant (Debio 1143) once daily from Day 1 to 14 per 3-week cycle in combination with with 66 Gray (Gy) of intensity modulated radiation therapy (IMRT) in 33 fractions, 2 Gy/fraction, 5 days/week followed by 3 cycles of monotherapy of placebo matched to Xevinapant (Debio 1143) from Day 1 to 14, per 3-week cycle (Each cycle is of 3 weeks).
  Interventions: Radiation: IMRT; Drug: Placebo

INTERVENTIONS:
Drug: Xevinapant — Participants received 3 cycles of oral solution of Xevinapant at a dose of 200 milligrams per day (mg/day) once daily from Day 1 to 14, per 3-week cycle.
  Other Names: Debio 1143
  Arms: Xevinapant + IMRT
Radiation: IMRT — Participants received 66 Gray (Gy) of intensity modulated radiation therapy (IMRT) in 33 fractions, 2 Gy/fraction, 5 days per week.
Drug: Placebo — Participants received 3 cycles of oral solution of placebo matched to Xevinapant once daily from Day 1 to 14 per 3-week cycle.
  Arms: Placebo + IMRT

SUMMARY:
The purpose of this study is to demonstrate the superior efficacy of Xevinapant (Debio 1143) versus placebo when added to radiotherapy in the treatment of high-risk participants with resected locally advanced squamous cell carcinoma of the head and neck (LA SCCHN) who are ineligible to receive cisplatin-based chemoradiation concurrently. Study details include: Study duration: Participants will be followed until the last on-study participant reaches his/her 60-month post-randomization visit, a decision to end the study has been triggered, or until premature discontinuation from study, whichever occurs first. Treatment duration: 18 weeks, consisting of six 3-week cycles. Health measurement/observation: Improved Disease-Free Survival. Visit frequency: Weekly visit during combination therapy period, once every 3 weeks during monotherapy period, and every 3, 4, or 6 months during the Disease-Free Survival Follow-up period in Year 1, 2 and 3, or 4 and 5 (with telephone contact in between), respectively, and every 3 months (telephone visits allowed) during the Overall Survival Follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-2 and able to tolerate standard of care IMRT treatment according to Investigator assessment
* Participants with histologically confirmed squamous cell carcinoma with one of the following primary sites: oral cavity, oropharynx, hypopharynx or larynx. Participants have received surgery with curative intent on these sites in the past 4 to 10 weeks before start of treatment (Cycle 1 Day 1)
* Oropharynx (OPC) participants must have known human papillomavirus (HPV) status as determined by p16 expression using immunohistochemistry (ICH)
* Participants with no residual disease by computed tomography (CT) or magnetic resonance imaging (MRI) and have a high risk of relapse with 1 or 2 of the following criteria, confirmed by local histopathology: • nodal extra-capsular extension (ECE) and positive resection margins (R1 or close margin less than or equal to (<=) 1 millimeter (mm)
* Are unfit to receive high-dose cisplatin by meeting one or more of the following criteria: estimated glomerular filtration rate (eGFR) < 60 milliliter per minute per 1.73 meter square (mL/min /1.73 m^2); History of hearing impairment, defined as Grade >= 2 audiometric hearing loss or tinnitus Grade >= 2. An audiogram is not required if one of the other criteria meets unfitness to receive high-dose cisplatin; Peripheral neuropathy > = Grade 2 and if >= 70 years, unfit according to G8 questionnaire (Score <= 14) or ineligible for cisplatin treatment due to age limit according to national guidelines
* Participants with adequate renal, hematologic and hepatic function as defined in the protocol
* Other protocol-defined inclusion criteria could apply

Exclusion Criteria:

* Any condition, including any uncontrolled disease state other than SCCHN that in the Investigator's opinion constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
* Participants with incomplete surgery
* Participants with recurrent or metastatic disease
* Primary tumor of nasopharyngeal, paranasal sinuses, nasal cavity, salivary, thyroid or parathyroid gland, skin or unknown primary site
* Prior definitive, neoadjuvant, concurrent or adjuvant (C)RT to the head and neck region which may jeopardize the primary tumor irradiation plan, or any other prior SCCHN systemic treatment, including investigational agents
* Participation in any interventional clinical study within 28 days prior to screening or during participation in this study
* Known contraindication to undergoing positron emission tomography with 18F-FDG-PET-CT scans, or both contrast-enhanced MRI and contrast-enhanced CT scans
* Known allergy to Xevinapant (Debio 1143) or any excipient known to be present in Xevinapant (Debio 1143) or in the placebo formulation
* Other protocol-defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | Time from randomization to the first occurrence of death from any cause or objective disease recurrence, assessed up to 5 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Time from randomization to death from any cause, assessed up to 5 years
Time to Subsequent Cancer Treatments | Time from randomization to the start of first subsequent cancer treatment, assessed up to 5 years
Number of Participants with Adverse Events (AEs) and Treatment-related AEs | Time from randomization until end of study (up to 5 years)
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Head and Neck Module (EORTC QLQ-HN35) Score | Baseline, Day 64 [at Week 10 (each cycle is 3 weeks)] and End of treatment Day 134 (at Week 20)
Change from Baseline in European Organization for research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30) Score | Baseline, Day 64 [at Week 10 (each cycle is 3 weeks)] and End of treatment Day 134 (at Week 20)
Change from Baseline in EuroQOL 5 Dimension 5 Level Health-Related Quality of Life Measure Visual Analog Scale Score (EQ-5D-5L VAS) | Baseline, Day 64 [at Week 10 (each cycle is 3 weeks)] and End of treatment Day 134 (at Week 20)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (206):
- United States (10):
  - University of Alabama at Birmingham - Dept of Radiation Oncology, Birmingham, Alabama
  - The University of Arizona Cancer Center, Tucson, Arizona
  - UC Health, Aurora, Colorado
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Perlmutter Cancer Center at NYU Langone Hospital ae Long Island, New York, New York
  - Montefiore Medical Center Radiology, The Bronx, New York
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - University of Pittsburgh Medical Center Health System - UPMC Department of Dermatology, Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute, ITOR, CRU, Greenville, South Carolina
- Argentina (5):
  - Instituto de Oncologia Angel Roffo, Ciudad Autonoma Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - CEMAIC- Centro Medico Privado, Las Margaritas
  - Fundacion Scherbovsky, Mendoza
  - Clinica Viedma S.A., Viedma
- Austria (3):
  - Universitatsklinikum Graz, Graz
  - Krankenhaus der barmherzigen Schwestern Linz - Abteilung für HNO, Linz
  - LKH - Universitätsklinikum der PMU Salzburg - Innere Med III/Hämatologie und Onkologie, Salzburg
- Belgium (4):
  - Institut Jules Bordet - Medical Oncology, Anderlecht
  - Cliniques Universitaires Saint-Luc - STL, Brussels
  - Antwerp University Hospital (UZA Parent), Edegem
  - Vitaz, Sint-Niklaas
- Brazil (16):
  - Hospital de Câncer de Barretos - Fundação Pio XII - Hospital de Amor, Barretos
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Câncer, Curitiba
  - CEPON - Centro de Pesquisas Oncológicas de Santa Catarina - Pesquisa Clínica, Florianópolis
  - CRIO - Centro Regional Integrado de Oncologia, Fortaleza
  - Oncosite - Centro de Pesquisa Clinica e Oncologia, Ijuí
  - Instituto de Cancer de Londrina, Londrina
  - Liga Norte-Rio-Grandense Contra o Câncer, Natal
  - HGB - Hospital Giovanni Battista - Mãe de Deus Center, Porto Alegre
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Grupo Oncoclínicas, Rio de Janeiro
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro
  - Hospital Santa Izabel - Santa Casa de Misericórdia da Bahia, Salvador
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia - Faculdade de Medicina do ABC, Santo André
  - BP A Beneficencia Portuguesa da Sao Paulo, São Paulo
  - ICESP - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira, São Paulo
- Centre Hospitalier de l'Universite de Montreal., Montreal, Canada
- China (25):
  - Beijing Cancer Hospital, Beijing
  - Hospital of Bengbu Medical College, Bengbu
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - Xiangya Hospital, Central South University, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Sir Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Anhui Provincial Cancer Hospital, Hefei
  - Shandong Cancer Hospital, Jinan
  - Jiangxi Cancer Hospital, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Union Hospital, Tongji Medical College of Huazhong University of Science & Technology, Wuhan
  - The Second Affiliated Hospital of Xi'an Jiaotong University（Xibei Hospital), Xi'an
  - Northern Jiangsu People's Hospital, Yangzhou
  - Henan Cancer Hospital, Zhengzhou
- Czechia (3):
  - Fakultni nemocnice Olomouc - Dept of Onkologicka klinika, Olomouc
  - Fakultni nemocnice Bulovka - Dept of Radiodiagnosticka klinika, Prague
  - Fakultni nemocnice Kralovske Vinohrady - Dept of Radioterapeuticka a onkologicka klinika, Prague
- France (25):
  - ICO - Site Paul Papin - service d'oncologie medicale, Angers
  - CHU Bordeaux - Service d'Oncologie Médicale, Bordeaux
  - CHU Brest - Hôpital Morvan - Service d'Oncologie Médicale, Brest
  - Centre Francois Baclesse - Service d'Oncologie Medicale, Caen
  - Centre Georges François Leclerc - Oncologie Médicale, Dijon
  - Hopital Prive Drome Ardeche - Service D Oncologie, Guilherand-Granges
  - Clinique Victor Hugo - Centre Jean Bernard - Service d'Oncologie Médicale, Le Mans
  - Centre Oscar Lambret - service de cancerologie gynecologique, Lille
  - Centre Hospitalier de Bretagne Sud, Lorient
  - Centre Hospitalier de la Croix Rousse - Service ORL et chirurgie cervico-faciale, Lyon
  - Hôpital de la Timone - Oncologie Médicale Hématologie & Soins Palliatifs, Marseille
  - Institut Régional du Cancer de Montpellier - Service de Professeur Senesse, Montpellier
  - Centre Azureen Cancerologie - Service De Radiotherapie, Mougins
  - Centre Antoine Lacassagne - Service d'Hématologie Oncologie, Nice
  - Hopital Tenon - service radiologie et imagerie medicale, Paris
  - Institut Curie - site de Paris - Service d'Oncologie Médicale, Paris
  - CHU Poitiers - Hôpital la Milétrie - service d'oncologie médicale, Poitiers
  - Centre Henri Becquerel - Service de radiothérapie, Rouen
  - Centre Hospitalier Privé Saint-Gregoire (Rennes) - Cancerologie, Saint-Grégoire
  - ICO - Site René Gauducheau - Service d'Oncologie medicale, Saint-Herblain
  - Institut de Cancérologie de Strasbourg Europe - ICANS - Service d'oncologie médicale, Strasbourg
  - CHI Toulon La Seyne - Hôpital Sainte Musse - Service d'Onco-Hematologie, Toulon
  - Institut Claudius Regaud - service de Radiothérapie, Toulouse
  - CHU Tours - Hôpital Bretonneau - Service d'Oncologie Médicale, Tours
  - Institut Gustave Roussy - Oncologie Médicale, Villejuif
- Georgia (6):
  - High Technology Hospital Medcenter LLC, Batumi
  - JSC EVEX Hospitals, Kutaisi
  - Cancer Research Center Ltd., Tbilisi
  - High Technology Medical Center, University Clinic, Tbilisi
  - LLC Todua Clinic, Tbilisi
  - New Hospitals, Tbilisi
- Germany (7):
  - Vivantes Klinikum Neukoelln - Parent, Berlin
  - Universitaetsklinikum Giessen und Marburg GmbH Standort Giessen - Hals-, Nasen- und Ohrenklinik, Giessen
  - Universitaetsmedizin Goettingen - Georg-August-Universität, Göttingen
  - Universitaetsklinikum Jena - HNO_Klinik, Jena
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel - Klinik für diagnostische Radiologie, Kiel
  - Universitaetsklinikum Leipzig - Klinik fuer Strahlentherapie und Radioonkologie, Leipzig
  - Universitaetsmedizin Rostock - Klinik und Poliklinik für Strahlentherapie, Rostock
- Greece (3):
  - General Hospital of Athens of Chest Diseases "SOTIRIA" - Sotiria Thoracic Diseases Hospital of Athens, Athens
  - University General Hospital "Attikon", Athens
  - Interbalkan Hospital of Thessaloniki, Thessaloniki
- India (4):
  - Tata Medical Centre, Kolkata
  - National Cancer Institute Nagpur, Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - Regional Cancer Centre, Thiruvananthapuram
- Israel (4):
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Chaim Sheba Medical Center - pt, Ramat Gan
- Italy (15):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili) - Oncologia Medica, Brescia
  - Ospedale Oncologico Armando Businco - Divisione di Oncologia Medica II, Cagliari
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo - Div. di Oncologia Medica ed Ematologia, Candiolo
  - Azienda Ospedaliera Universitaria Careggi - S.O.D. di Oncologia Medica, Florence
  - IRCCS Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori "Dino Amadori" - IRST - U. Operativa di Immunoterapia e Terapia Cellulare, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori - S.S. Tumori della Testa e del Collo, Milan
  - IEO Istituto Europeo di Oncologia - Divisione Oncologia Medica, Milan
  - Ospedale San Raffaele - U.O. di Oncologia Medica, Milan
  - A.O.U. Policlinico di Modena - U.O. Oncologia, Modena
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania "Luigi Vanvitelli" - Dipartimento Oncologia, Napoli
  - Istituto Nazionale Tumori Fondazione G. Pascale - Oncologia Medica A, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS - Oncologia Medica 2, Padua
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza - U.O.C. di Oncologia B, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Radioterapia 1, Roma
  - Istituto Clinico Humanitas - U.O. di Oncologia Medica ed Ematologia, Rozzano
- Japan (20):
  - Hyogo Cancer Center - Dept of Head and Neck Surgery, Akashi-shi
  - National Cancer Center Hospital - Dept of Gastroenterology, Chūōku
  - NHO Kyushu Cancer Center - Dept of Head and Neck Surgery, Fukuoka
  - Saitama Medical University International Medical Center - Dept of Otorhinolaryngology/ Head and Neck Surgery, Hidaka-shi
  - Hiroshima University Hospital - Dept of Otorhinolaryngology/ Head and Neck Surgery, Hiroshima
  - National Cancer Center Hospital East - Dept of Head and Neck Medical Oncology, Kashiwa-shi
  - Kagawa University Hospital - Dept of Oncology, Kita-gun
  - Saitama Cancer Center - Dept of Head and Neck Surgery, Kitaadachi-gun
  - Kobe University Hospital - Dept of Oncology/Hematology, Kobe
  - Cancer Institute Hospital of JFCR - Dept of Medical Oncology, Kōtoku
  - NHO Shikoku Cancer Center - Dept of Head and Neck Surgery, Matsuyama
  - Aichi Cancer Center Hospital - Dept of Head and Neck Surgery, Nagoya
  - Nagoya University Hospital - Dept of Otorhinolaryngology, Nagoya
  - Okayama University Hospital - Dept of Otorhinolaryngology, Okayama
  - Osaka International Cancer Institute - Dept of Head and Neck Surgery, Osaka
  - Kindai University Hospital - Dept of Oncology, Osakasayama-shi
  - Hokkaido University Hospital - Dept of Otorhinolaryngology, Sapporo
  - NHO Hokkaido Cancer Center - Dept of Oral Oncology Surgery, Sapporo
  - Tohoku University Hospital - Dept of Otorhinolaryngology/Head and Neck Surgery, Sendai
  - Yokohama City University Hospital - Dept of Otorhinolaryngology, Yokohama
- Mexico (3):
  - Hospital Civil Fray Antonio Alcalde - O.P.D. Hospital Civil de Guadalajara, Guadalajara
  - Centro de Atención e Investigación Clínica en Oncología, Mérida
  - Universidad Autonoma de Nuevo Leon, Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey
- Netherlands (3):
  - Amsterdam UMC, Locatie VUMC - Dept of Medical Oncology, Amsterdam
  - Universitair Medisch Centrum Groningen - Cancer Center, Groningen
  - UMC Utrecht - Dept Medical Oncology, Utrecht
- Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie, Państwowy Instytut Badawczy - Zakład Medycyny Nuklearnej i Endokrynologii Onkolo, Gliwice, Poland
- Portugal (2):
  - Hospital de Braga - Serviço de Oncologia Medica, Braga
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
- Romania (5):
  - Centrul medical Focus, Bucharest
  - S.C Medisprof S.R.L - parent, Cluj-Napoca
  - S.C Radiotherapy Center Cluj S.R.L - Parent, ComunaFloresti
  - S.C Centrul de Oncologie Sf. Nectarie S.R.L - parent, Craiova
  - S.C Oncocenter Oncologie Clinica S.R.L - parent, Timișoara
- South Korea (6):
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Seoul National University Bundang Hospital, Seongnam
  - Konkuk University Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (14):
  - Complejo Hospitalario Universitario A Coruña - CHUAC-Hospital Teresa Herrera, A Coruña
  - Complejo Hospitalario Universitario A Coruña - Servicio de Oncologia, A Coruña
  - Hospital Clinic de Barcelona - Medical Oncology, Barcelona
  - Hospital del Mar - Servicio de Oncologia, Barcelona
  - Hospital Universitari Vall d'Hebron - Oncology Dept., Barcelona
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol - Servicio de Oncologia Medica, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals - Servicio de Oncologia, Barcelona
  - Complejo Hospitalario Universitario Insular Materno-Infantil - Servicio de Oncologia, Las Palmas de Gran Canaria
  - Hospital Universitario Lucus Augusti - Oncology, Lugo
  - Clinica Universidad de Navarra (MAD) - Oncology Service, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz - Oncology, Madrid
  - Hospital Universitario La Paz - Oncology Department, Madrid
  - Hospital Regional Universitario de Malaga - Oncology Dept, Málaga
  - Hospital Universitario Virgen del Rocio - Oncology Service, Seville
- Switzerland (4):
  - Universitaetsspital Basel - Klinik fuer Strahlentherapie und Radioonkologie, Basel
  - Istituto Oncologico della Svizzera Italiana (IOSI)- Ente Ospedaliero Cantonale (EOC) - Ospedale S.Giovanni, Bellinzona
  - CHUV, Lausanne University Hospital, Lausanne
  - Universitaetsspital Zuerich - Parent, Zurich
- Taiwan (9):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chi Mei Hospital, Liouying, Tainan
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital,Linkou, Taoyuan District
- United Kingdom (8):
  - St James's University Hospital - Dept of Oncology, Leeds
  - Royal Marsden Hospital-London - Dept of Haematology/Oncology Research, London
  - The Christie Hospital - Dept of Oncology, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Mount Vernon Cancer Centre, Northwood
  - Musgrove Park Hospital - PARENT, Somerset
  - The Royal Marsden NHS Foundation Trust, Sutton
  - Torbay Hospital - PARENT, Torquay

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Derived] Ferris RL, Mehanna H, Schoenfeld JD, Tahara M, Yom SS, Haddad R, Konig A, Witzler P, Bajars M, Tourneau CL. Xevinapant plus radiotherapy in resected, high-risk, cisplatin-ineligible LA SCCHN: the phase III XRay Vision study design. Future Oncol. 2024 Apr;20(12):739-748. doi: 10.2217/fon-2023-0774. Epub 2024 Jan 10. PMID 38197296
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS202359_0002
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html